CLINICAL TRIAL: NCT06054243
Title: Efficacy of Group Cognitive Behavioural Therapy for Youth Anxiety and Insomnia: A Randomised, Assessor Blind, Parallel-group Trial
Brief Title: Efficacy of Group Cognitive Behavioural Therapy for Youth Anxiety and Insomnia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Chinese University of Hong Kong (Other); Goldsmiths, University of London (Other); Stanford University (Other)
Responsible Party: Principal Investigator, Dr. Shirley Xin Li, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EA210509
Record Dates: First submitted 2023-09-19; First posted 2023-09-26 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Insomnia; Anxiety
Keywords: Insomnia; Anxiety; Adolescents; Youth
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CBT-I (Experimental)
  Interventions: Behavioral: CBT-I
- CBT-A (Active Comparator)
  Interventions: Behavioral: CBT-A
- Waiting-list control (No Intervention)

INTERVENTIONS:
Behavioral: CBT-I — The intervention will consist of eight weekly group sessions (120-min, 5-8 adolescents in each group) delivered within a 10-week windows. The treatment components aim to address the behavioural, cognitive and physiological factors perpetuating insomnia whilst considering the sleep and circadian features in adolescents and developmental context with the following key elements: psychoeducation about sleep, circadian rhythm and sleep hygiene, stimulus control, sleep restriction, relaxation training, structured worry time, cognitive restructuring (targeting sleep-related dysfunctional cognitions), and relapse prevention.
  Arms: CBT-I
Behavioral: CBT-A — The intervention will consist of eight weekly group sessions (120-min, 5-8 adolescents in each group) delivered within a 10-week windows. The CBT-A treatment is modified from the Coping Cat programme, which incorporates psychoeducation and the core behavioural strategies and cognitive skills for managing anxiety (e.g. exposure, relaxation training, cognitive restructuring).
  Arms: CBT-A

SUMMARY:
Youth is an important transitional stage associated with dynamic changes in biological, cognitive, and psychological functioning, as well as a constellation of developmental and psychosocial challenges. In particular, anxiety disorders constitute the most common mental health problems in youth, with a prevalence rate up to 32%. Youth anxiety is associated with not only profound personal distress, but also considerable impairments in psychosocial functioning and an increased risk for developing other psychiatric comorbidities (e.g. depression, substance use). Meanwhile, sleep problems, particularly insomnia, are also common in the teen years, with a prevalence rate as high as 36%. Insomnia and anxiety are highly comorbid conditions, with increasing evidence suggesting their intricate, bidirectional relationship, such as a high level of anxiety symptoms found in youth with insomnia. However, optimal treatment strategies to manage the comorbidity of these two conditions remain uncertain. This study will test the efficacy of group-based cognitive behavioural therapy for insomnia (CBT-I) and cognitive behavioural therapy for anxiety (CBT-A) in reducing the severity of insomnia and anxiety symptoms in youth with comorbid insomnia and anxiety, as well as their effects on depressive symptoms, daytime functioning (e.g. sleepiness, fatigue), subjective and objective sleep measures.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese aged 12-20 years old (an age range that was suggested by scholars to cover a wider developmental span in adolescence);
2. Written informed consent of participation into the study is given by the participant and his/her parent or guardian (for those aged under 18);
3. Willing to comply with the study protocol;
4. Meeting the DSM-5 diagnostic criteria of insomnia disorder and with a score on Insomnia Severity Index (ISI) >= 9 (suggested cut-off for adolescents); 5) Presenting with a high level of anxiety symptoms as defined by a total score >32 and >37 for males and females respectively on Spence Children's Anxiety Scale (SCAS).

Exclusion Criteria:

1. A current diagnosis of substance abuse or dependence; a current or past history of manic or hypomanic episode, schizophrenia spectrum disorders, neurodevelopmental disorders, organic mental disorders, or intellectual disabilities;
2. Having a prominent medical condition known to interfere with sleep continuity and quality (e.g. eczema, gastro-oesophageal reflux disease);
3. Having a clinically diagnosed sleep disorder (other than insomnia) that may potentially contribute to a disruption in sleep continuity and quality, such as narcolepsy, sleep-disordered breathing, and restless leg syndrome, as ascertained by the DISP, a validated structured diagnostic interview to assess major sleep disorders according to the ICSD criteria;
4. Concurrent, regular use of medications(s) known to affect sleep continuity and quality including both western medications (e.g. hypnotics, steroids) and over-the-counter OTC medications (e.g. melatonin, Traditional Chinese Medicine, TCM);
5. Having been enrolled in any other clinical trial investigational products within one month at the entry of the study;
6. Having a clinically significant suicidality (presence of suicidal ideation with a plan or an attempt) as assessed confirmed by research clinician using the MINI Suicidality Module;
7. Currently receiving any structured psychotherapy;
8. With hearing or speech deficit;
9. Night shift worker.

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 171 (Estimated)
Dates: Start 2023-02-17 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change of anxiety symptoms (assessor-rated) | Baseline, post-treatment (one-week after completion of the intervention/waiting period) for all participants; and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  Pediatric Anxiety Rating Scale (PARS) is a clinician-rated scale commonly used in the clinical studies on anxiety conducted in adolescents. Possible scores range from 0 to 35, with higher scores indicating severer anxiety symptoms.
Change of insomnia symptoms | Baseline, post-treatment (one-week after completion of the intervention/waiting period) for all participants; and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  Insomnia Severity Index (ISI) is a 7-item self-rated scale. Possible scores range from 0 to 20, with higher scores indicating greater insomnia severity.

SECONDARY OUTCOMES:
Change of sleep quality | Baseline, post-treatment (one-week after completion of the intervention/waiting period) for all participants; and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  Pittsburgh Sleep Quality Index (PSQI) is a self-rated scale consisting of 19 questions. All items are combined to form seven component scores on different aspects of sleep quality, each of which ranges from 0 to 3 points with higher scores representing more sleep disturbance. The seven component scores are added to one global score, which ranges from 0 to 21, with higher scores indicating more difficulties with sleep.
Change of sleep diary measure (time in bed, TIB) | Baseline, post-treatment (one-week after completion of the intervention/waiting period) for all participants; and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  Daily sleep diary for consecutive seven days. Sleep parameter estimated by daily sleep diary: time in bed (TIB) in hours
Change of sleep diary measure (total sleep time, TST) | Baseline, post-treatment (one-week after completion of the intervention/waiting period) for all participants; and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  Daily sleep diary for consecutive seven days. Sleep parameter estimated by daily sleep diary: time in bed (TIB) in hours
Change of sleep diary measure (sleep onset latency, SOL) | Baseline, post-treatment (one-week after completion of the intervention/waiting period) for all participants; and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  Daily sleep diary for consecutive seven days. Sleep parameter estimated by daily sleep diary: total sleep time (TST) in hours
Change of sleep diary measure (wake after sleep onset, WASO) | Baseline, post-treatment (one-week after completion of the intervention/waiting period) for all participants; and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  Daily sleep diary for consecutive seven days. Sleep parameter estimated by daily sleep diary: wake after sleep onset (WASO) in mins
Change of sleep diary measure (sleep efficiency, SE) | Baseline, post-treatment (one-week after completion of the intervention/waiting period) for all participants; and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  Daily sleep diary for consecutive seven days. Sleep parameter estimated by daily sleep diary: sleep efficiency (SE), which is calculated by total sleep time divided by total time in bed, %
Change of objective sleep measure (time in bed, TIB) | Baseline, post-treatment (one-week after completion of the intervention/waiting period) for all participants; and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  Actigraphic assessment for consecutive seven days. Sleep parameter estimated by wrist actigraphy: time in bed (TIB) in hours
Change of objective sleep measure (total sleep time, TST) | Baseline, post-treatment (one-week after completion of the intervention/waiting period) for all participants; and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  Actigraphic assessment for consecutive seven days. Sleep parameter estimated by wrist actigraphy: total sleep time (TST) in hours
Change of objective sleep measure (sleep onset latency, SOL) | Baseline, post-treatment (one-week after completion of the intervention/waiting period) for all participants; and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  Actigraphic assessment for consecutive seven days. Sleep parameter estimated by wrist actigraphy: sleep onset latency (SOL) in mins
Change of objective sleep measure (wake after sleep onset, WASO) | Baseline, post-treatment (one-week after completion of the intervention/waiting period) for all participants; and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  Actigraphic assessment for consecutive seven days. Sleep parameter estimated by wrist actigraphy: wake after sleep onset (WASO) in mins
Change of objective sleep measure (sleep efficiency, SE) | Baseline, post-treatment (one-week after completion of the intervention/waiting period) for all participants; and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  Actigraphic assessment for consecutive seven days. Sleep parameter estimated by wrist actigraphy: sleep efficiency (SE), which is calculated by total sleep time divided by total time in bed, %
Change of dysfunctional beliefs and attitudes about sleep | Baseline, post-treatment (one-week after completion of the intervention/waiting period) for all participants; and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  Dysfunctional Beliefs and Attitudes about Sleep (DBAS) is a 16-item self-rated scale measuring the respondent's sleep-related beliefs, more specifically, their expectations and attitudes regarding the causes, consequences, and potential treatments of sleep issues. A total score is calculated by averaging score of all items, possibly scored 0 to 10, with a higher score indicating more dysfunctional beliefs and attitudes about sleep.
Change of pre-sleep arousal | Baseline, post-treatment (one-week after completion of the intervention/waiting period) for all participants; and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  Pre-Sleep Arousal Scale is a 16-item self-rated scale measuring pre-sleep arousal. There are two subscales on the cognitive and somatic manifestations of arousal, with eight items in each subscale (possibly scored from 8 to 40). In both cases, a higher score indicates higher pre-sleep arousal.
Change of sleep reactivity | Baseline, post-treatment (one-week after completion of the intervention/waiting period) for all participants; and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  Ford Insomnia Response to Stress Test (FIRST) is a 9-item self-rated scale measuring sleep reactivity. Possible scores range from 9 to 36. A higher score indicates higher sleep activity.
Change of sleep hygiene and practice | Baseline, post-treatment (one-week after completion of the intervention/waiting period) for all participants; and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  Sleep Hygiene Practice Scale (SHPS) is a 30-item self-rated scale measuring sleep hygiene behaviors, ranging in total scores from 30 to 180, with higher scores indicating lower levels of sleep hygiene.
Change of daytime sleepiness | Baseline, post-treatment (one-week after completion of the intervention/waiting period) for all participants; and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  Paediatric Daytime Sleepiness Scale (PDSS) is an 8-item self-rated scale measuring daytime sleepiness, ranging in total scores from 0 to 32 with higher scores indicating more sleepiness.
Change of daytime hyperarousal | Baseline, post-treatment (one-week after completion of the intervention/waiting period) for all participants; and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  Hyperarousal Scale (HAS) is a 26-item self-rated scale measuring arousal and alertness during wakefulness. Possible total scores range from 0 to 78, with higher scores indicating higher hyperarousal.
Change of daytime fatigue | Baseline, post-treatment (one-week after completion of the intervention/waiting period) for all participants; and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  Multidimensional Fatigue Inventory (MFI) is a 20-item self-rated scale on fatigue symptoms. There are three subscales, measuring the physical (possibly scored from 7 to 35), mental (possibly scored from 6 to 30), and spiritual (possibly scored from 7 to 35), dimensions of fatigue. A grand total score can be calculated by summing up the three sub scores. In all cases, a higher score represents higher fatigue symptoms.
Change in sleep timing and chronotype | Baseline, post-treatment (one-week after completion of the intervention/waiting period) for all participants; and additional one follow-up at Post-Treatment 6-month for participants in the treatment groups
  The Munich Chronotype Questionnaire (MCTQ) is a 14-item self-rated scale measuring sleep patterns during weekdays and weekends separately. The Mid-Sleep Time (MSF/MSFsc) are used to as an indicator of chronotype, where individuals with earlier mid-sleep time reflect a morning chronotype and later mid-sleep time reflect an evening chronotype.
Change in chronotype preference | Baseline, post-treatment (one-week after completion of the intervention/waiting period) for all participants; and additional one follow-up at Post-Treatment 6-month for participants in the treatment groups
  The Morningness-Eveningness Questionnaire (MEQ) is a 19-item self-rated scale measuring chronotype preference. Possible total scores range from 16 to 86, with higher scores indicating morningness and lower scores indicating eveningness.
Change in anxiety symptoms | Baseline, post-treatment (one-week after completion of the intervention/waiting period) for all participants; and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  The Spence Children's Anxiety Scale (SCAS) is a 44-item self-rated scale measuring six types of anxiety symptoms in children and adolescents, with 6 positive filler items. Possible total scores range from 0 to 114, with higher scores indicating more anxiety symptoms.
Change of mood symptoms | Baseline, post-treatment (one-week after completion of the intervention/waiting period) for all participants; and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  The Hospital Anxiety and Depression Scale (HADS) is a self-assessed scale for detecting states of depression and anxiety. The depression subscale range in scores from 0 to 21, with higher scores indicating severer states of depression. Similarly, the anxiety subscale range in scores from 0-21 with higher scores indicating severer states of anxiety. No additional computation will be made with the two subscores.
Change of emotional states of depression, anxiety, and stress | Baseline, post-treatment (one-week after completion of the intervention/waiting period) for all participants; and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  The Depression Anxiety Stress Scales (DASS-21) is a 42-item self-rated scale measuring the emotional states of depression, anxiety and stress, with three subscales. Higher scores suggest more depression, anxiety, and stress, respectively.
Change of suicidal ideation | Baseline, post-treatment (one-week after completion of the intervention/waiting period) for all participants; and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  The Depressive Symptom Inventory Suicidality Subscale (DSI-SS) is a 4-item self-rated scale measuring suicidal ideation. Possible total scores range from 0 to 12, with higher scores indicating higher suicidal ideation.
Change of state and trait anxiety | Baseline, post-treatment (one-week after completion of the intervention/waiting period) for all participants; and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  The State-Trait Anxiety Inventory (STAI) is a 40-item self-rated scale measuring the intensity of state and trait anxiety, divided into two subscales of 20 items per each. Higher scores suggest higher state and trait anxiety.
Change of Locus of Control | Baseline, post-treatment (one-week after completion of the intervention/waiting period) for all participants
  The Locus of Control Scale (LCS) is a 29-item scale measuring an individual's locus of control. A higher score indicates externally oriented, while a lower score indicates internally oriented.
Change of Sleep-related Locus of Control | Baseline, post-treatment (one-week after completion of the intervention/waiting period) for all participants
  The Sleep Locus of Control Scale (SLOCS) is an 8-item questionnaire measuring sleep-related locus of control. It is represented by two dimensions, including "internal sleep locus" and "chance sleep locus," with a 6-point scale ranging from 1 (strongly disagree) to 6 (strongly agree).
Change of Repetitive Negative Thinking | Baseline, post-treatment (one-week after completion of the intervention/waiting period) for all participants
  The Perseverative Thinking Questionnaire is a 15-items scale measuring repetitive negative thinking. It comprised 5 assumed process characteristics of repetitive negative thinking, with three items per each characteristics. Each item is rated on a 5-point Likert Scale ranging from never to almost always.
Change of quality of life | Baseline, post-treatment (one-week after completion of the intervention/waiting period) for all participants; and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  KIDSCREEN-27 is a 27-item self-rated scale measuring health related quality of life measure for children and adolescents. There are five subscales on: physical well-being (possibly scored from 5 to 25), psychological well-being (possibly scored 7 to 35), autonomy & parents (possibly scored 7 to 35), peers & social support (possibly scored 4 to 20), and school environment (possibly scored 4 to 20). A grand total score can be calculated by summing up the five sub scores. In all cases, a higher score represents higher perceived well-being.
Change of overall severity of clinical symptoms | Baseline, post-treatment (one-week after completion of the intervention/waiting period) for all participants; and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  Clinical Global Impression (CGI) Scale is a clinician-rated scale, comprised of two one-item subscales: Severity of Illness (CGI-S) subscale evaluating the severity of psychopathology, and Clinical Global Improvement Scale (CGI-I) evaluating change from the initiation of treatment. In both cases, the score is given on a seven-point scale, with higher values indicating higher severity of illness and larger improvement respectively.
Change of objective cognitive performance (attentional bias) | Baseline, post-treatment (one-week after completion of the intervention/waiting period) for all participants; and additional one follow-up at Post-Treatment 6-month for participants in the treatment groups
  Threat- and Sleep-related Dot-probe Task for assessing attentional bias, where an attentional bias interference score will be computed based on the response time to congruent and incongruent trials. A positive score indicates vigilance to threat whilst a negative score indicates avoidance.
Change of objective physiological performance (attentional bias) | Baseline, post-treatment (one-week after completion of the intervention/waiting period) for all participants; and additional one follow-up at Post-Treatment 6-month for participants in the treatment groups
  Additional eye-tracking measure on Threat- and Sleep-related Dot-probe Task for assessing attentional bias. Specific eye-gaze patterns will be estimated by a Hidden Markov Models (EMHMM).
Change of objective cognitive performance (working memory) | Baseline, post-treatment (one-week after completion of the intervention/waiting period) for all participants; and additional one follow-up at Post-Treatment 6-month for participants in the treatment groups
  N-back Task for assessing working memory capacity and manipulation. In N-back Task, a d prime score will be calculated based on the signal detection theory, where a higher score indicates better working memory performance.
Change of objective cognitive performance (working memory) | Baseline, post-treatment (one-week after completion of the intervention/waiting period) for all participants; and additional one follow-up at Post-Treatment 6-month for participants in the treatment groups
  Digit Span Task for assessing working memory capacity. In Digit Span Task, a higher number of recalled digits indicates better working memory.
Change of objective cognitive performance (inhibitory ability) | Baseline, post-treatment (one-week after completion of the intervention/waiting period) for all participants; and additional one follow-up at Post-Treatment 6-month for participants in the treatment groups
  Go/No-go Task for assessing inhibitory ability. In Go/No-go Task, a higher error rate indicates lower inhibition control.
Change of objective cognitive performance (risk-taking & decision making) | Baseline, post-treatment (one-week after completion of the intervention/waiting period) for all participants; and additional one follow-up at Post-Treatment 6-month for participants in the treatment groups
  Balloon Analogue Risk Task for assessing risk-taking and decision-making. In Balloon Analogue Risk Task, a score will be calculated by averaging the number of pumps on unexploded blue balloons, where a higher score indicates more risk-taking and impulsive propensities.

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Xin Li, PhD, DClinPsy, Principal Investigator — The University of Hong Kong
Locations (1):
- Sleep Research Clinic & Laboratory, Department of Psychology, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No